CLINICAL TRIAL: NCT05898919
Title: Acupuncture Versus Sham Acupuncture and Neostigmine for the Management of Postoperative Urinary Retention
Brief Title: Acupuncture for Postoperative Urinary Retention After Hemorrhoidectomy: a Randomized Controlled Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Hui Zheng, Clinical Professor, Chengdu University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HCDUTCM_2022056
Record Dates: First submitted 2023-05-27; First posted 2023-06-12 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Postoperative Complications; Postoperative Urinary Retention
MeSH Terms: conditions — Postoperative Complications | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupuncture (Experimental)
  Interventions: Other: Acupuncture
- Sham acupuncture (Placebo Comparator)
  Interventions: Other: Sham acupuncture
- Neostigmine (Active Comparator)
  Interventions: Drug: Neostigmine Injectable Product

INTERVENTIONS:
Other: Acupuncture — Acupuncture is a technique that inserts a needle into the acupuncture point to treat a condition. In this trial, we will use acupuncture to treat postoperative urinary retention.
  Arms: Acupuncture
Other: Sham acupuncture — Participants will receive sham acupuncture at sham points.
  Arms: Sham acupuncture
Drug: Neostigmine Injectable Product — Neostigmine was injected once after postoperative urinary retention.
  Arms: Neostigmine

SUMMARY:
The goal of this study is to examine the efficacy of acupuncture in the management of acute postoperative urinary retention.

Clinical question:

Is acupuncture efficacious for postoperative urinary retention after hemorrhoidectomy compared with sham acupuncture and neostigmine.

Study design:

The participants who undergo hemorrhoidectomy and report postoperative urinary retention will receive one session of acupuncture or sham acupuncture or one injection of 1-mg neostigmine. The primary outcome was the time to first urination after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years
* Meets the diagnostic criteria of postoperative urinary retention
* Received milligan-morgan hemorrhoidectomy and general anesthesia

Exclusion Criteria:

* Received Diuretic drugs
* Organic diseases that cause urinary retention
* Severe infection in the urinary tract
* Has a history of adverse reaction to neostigmine
* Cognitive dysfunction that affects outcome assessment
* Being pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-07-06 (Actual)

PRIMARY OUTCOMES:
The time to first urination after surgery | Immediately after first urination
  This outcome records the time period from the end of surgery to the immediately first urination.

SECONDARY OUTCOMES:
The volume of first of urination | Immediately after first urination
  This outcome measures the total volume of the first urination after surgery.
Bladder residual urine volume | 10 minutes before treatment, 0.5, 1, and 2 hours after treatment.
  This outcome measures the bladder residual urine volume using the ultrasound measurement.
Urination Score | 10 minutes before treatment, 0.5, 1, and 2 hours after treatment.
  The urination score ranges from 0 to 4 points. A higher score indicates more difficult to urinate.
Abdominal symptom score | Before treatment, 0.5, 1, and 2 hours after treatment.
  The abdominal symptom score ranges from 0 to 3 points. A higher score indicates worse abdominal symptoms.
Visual analogue score after surgery | 2 hours after treatment.
  The visual analogue score ranges from 0 to 10 cm. A higher score indicates more painful symptoms.
Adverse effects | 48 hours after treatment
  The adverse events will recorded by the patients and evaluated by the physicians. And the adverse events will be classified into mild and severe. Mild adverse events need no additional medical care.

CONTACTS AND LOCATIONS:
Overall Officials: Min Chen, MD, Principal Investigator — Chengdu University of Traditional Chinese Medicine
Locations (1):
- Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu, China

IPD SHARING:
Plan to Share IPD: Undecided